CLINICAL TRIAL: NCT02054728
Title: Inspiratory Muscle Training During Right-heart Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: WI_IMT_RHK_82/2012
Record Dates: First submitted 2012-12-20; First posted 2014-02-04 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Right-heart Hemodynamics; Respiratory Muscle Training; Inspiratory Resistance
Keywords: right-heart catheterization; respiratory muscle training; inspiratory resistance; hemodynamics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RHC and IMT (Experimental)
  Interventions: Other: RHC and IMT

INTERVENTIONS:
Other: RHC and IMT — Eligible patients subjected to RHC will be instructed on how to do RMT using the Threshold IMT® two days in advance. RMT will be conducted with 20-30% of individual inspiratory muscle strength, which will be measured beforehand. A single training session consists of 7 cycles with 2 min inspiratory training each, followed by a 1 min break (total duration 21 min).
  The actual intervention consists of inspiratory muscle training (IMT) during right-heart catheterization for at least 2 min or as long as is necessary to measure all specified parameters.

SUMMARY:
The purpose of this study is to assess hemodynamic effects of inspiratory muscle training during routinely performed right-heart catheterization.

DETAILED DESCRIPTION:
During the last years, respiratory muscle training (RMT) in patients with impaired respiratory muscle function, e.g. in chronic obstructive pulmonary disease (COPD), is increasingly applied. RMT can be done by applying increased respiratory effort for several minutes via an apparatus providing an inspiratory stenosis. Threshold IMT® (Philips Respironics) for example is such a training device, which is in the market for several years now and which has been used to conduct studies applying RMT. For example, it has been shown that training with the Threshold IMT® in patients with COPD increases inspiratory muscle strength, endurance and functional capacity and ameliorates dyspnea and quality of life. Furthermore, patients suffering from cardiac illness can also be affected by respiratory muscle impairment, which can add to their cardiogenic dyspnea. RMT can help improve dyspnea and physical exercise capacity in those patients as well.

To date, no studies have been performed addressing acute hemodynamic effects of inspiratory muscle training. However, this is of special interest: COPD as well as heart failure patients show an increased prevalence of pulmonary hypertension.

In case of suspected pulmonary hypertension, patients usually are subjected to right-heart catheterization (RHC) to arrive at a definitive diagnosis and assess severity and etiology of potentially present pulmonary hypertension. RHC is also a sensitive method to exclude an intracardial shunt in COPD patients.

In this study, patients who are routinely subjected to RHC for the above mentioned reasons will be instructed to do RMT using the Threshold IMT® during RHC. Two days in advance they will begin a guided training to get familiar with the Threshold IMT®. The device's inspiratory resistance can be set between 9 and 41 cm H2O. A single training session consists of 7 cycles with 2 min inspiratory training each, followed by a 1 min break (total duration 21 min). RMT will be conducted with 20-30% of individual inspiratory muscle strength, which will be measured beforehand.

During the RHC procedure the patients will again conduct RMT as instructed while the suspected hemodynamic effects will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Indication for right-heart catheterization
* Informed Consent provided

Exclusion Criteria:

* Age < 18 years
* Inability or contraindication to undergo right-heart catheterization
* Inability or contraindication to undergo respiratory muscle training as required per protocol
* Pregnancy, lactation
* Any medical, psychological or other condition restricting the patient's ability to provide informed consent
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10-16 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2014-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Pulmonary arterial pressure | During RHC with and without parallel IMT
  Pulmonary arterial pressure will be measured during RHC with and without parallel Inspiratory Muscle Training (IMT). Changes related to IMT will be assessed.

SECONDARY OUTCOMES:
Change in Pulmonary Capillary Wedge Pressure | During RHC with and without parallel IMT
Change in Cardiac output | During RHC with and without parallel IMT
Change in Cardiac index | During RHC with and without parallel IMT
Change in Stroke volume index | During RHC with and without parallel IMT
Change in Stroke volume | During RHC with and without parallel IMT

CONTACTS AND LOCATIONS:
Locations (1):
- Bethanien Hospital, Clinic for Pneumology and Allergology, Center for Sleep and Respiratory Medicine, Solingen, North Rhine-Westphalia, Germany